CLINICAL TRIAL: NCT04276974
Title: Effects of an Organic Plant-rich Diet on Gut Microbiome and Vascular Function: the ORGAMIC Pilot Study
Brief Title: Effects of an Organic Plant-rich Diet on Gut Microbiome and Vascular Function (ORGAMIC Pilot Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Ana Rodriguez-Mateos, Principal Investigator, Lecturer in Nutritional Sciences, King's College London
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HR-19/20-14
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Healthy Men and Women
Keywords: polyphenols; pesticides; plant based food; organic; microbiome; vascular function

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Organic first then non-organic (Experimental): Organic diet then non-organic diet, each for 4 consecutive days
  Interventions: Other: Organic diet; Other: Non-organic diet
- Non-organic first then organic (Experimental): Non-organic diet then organic diet, each for 4 consecutive days
  Interventions: Other: Organic diet; Other: Non-organic diet

INTERVENTIONS:
Other: Organic diet — Organic plant-rich foods (2000kcal for women, 2500kcal for men)
Other: Non-organic diet — Likewise Non-organic plant-rich foods (2000kcal for women, 2500kcal for men)

SUMMARY:
Previous work have shown that consumption of foods rich in polyphenols, such as berries and cocoa, led to beneficial changes in the gut microbiota composition, as well as improvements in biomarkers of cardiovascular disease risk in healthy volunteers. In addition, recent studies suggest that pesticide exposure has a detrimental effect on the gut microbiome in human populations and laboratory animals.The aim of this pilot study is to investigate the effects of short-term consumption of an organic and a non-organic plant rich diet on urinary polyphenol and pesticide levels, gut microbiome and selected biomarkers of cardiovascular health in a group of young healthy individuals.

Healthy men and women participants (10) will be recruited for a 2-arm randomised crossover controlled trial. Urinary polyphenol and pesticide levels after consumption of an organic and non-organic plant rich diet for 4 days will be analysed. Changes in gut microbiome composition and biomarkers of cardiovascular disease risk (flow-mediated dilation, blood pressure and arterial stiffness) will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 20-40 years old.
* Body mass index between 18.5 and 30 kg/m2.
* Non-smokers
* Not already participating in a clinical trial.
* No diagnosed heart attack, stroke, angina, thrombosis, liver or kidney diseases, diabetes, chronic gastrointestinal disorder or cancer.
* Not currently taking any medication
* No history of excess alcohol intake or substance abuse.
* Happy to follow dietary instructions before and during the study and to attend the research centre for breakfast and lunch for a total of 10 days.
* Ability to prepare basic meals from ingredients provided.
* No food intolerances, allergies, hypersensitivity or follow any dietary restriction (e.g. gluten intolerance, coeliac, lactose intolerance) that will prevent your ability to follow the test diets.
* Weight stable (no weight change by more than 3 kg in the last 2 months).
* No travel arrangements outside the United Kingdom (UK) within the period of data collection.
* Able to understand the information sheet and willing to comply with study protocol.
* Able to give informed written consent.

Exclusion Criteria:

* Women who are pregnant, intending to become pregnant, or breastfeeding.
* Participation in another clinical trial - Unable to comply with the study protocol.
* Weight change >3kg in preceding 2 months and body mass index <18.5 or >30 kg/m2
* Current smokers, or reported giving up smoking within the last 6 months History of substance abuse, previous or current high alcohol intake (>28 units/week for males and >21 units/week for females).
* Reported history of Cardiovascular disease, diabetes, cancer, kidney, liver or bowel disease, gastrointestinal disorder or use of drug likely to alter gastrointestinal function)
* Blood pressure ≥160/100 mmHg
* Travel arrangements outside UK within the period of data collection.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-07-17 (Actual)

PRIMARY OUTCOMES:
Changes in urinary pesticides levels | Baseline & 4 days after
  Determine changes in urinary pesticides levels after consumption of organic plant-rich diet for 4 days measuring by chromatography coupled with mass spectrometry analytical techniques (HPLC-MS)
Changes in urinary polyphenol levels | Baseline & 4 days after
  Determine changes in urinary polyphenol profiles after consumption of organic or non-organic plant-rich diet for 4 days measuring by chromatography coupled with mass spectrometry analytical techniques (HPLC-MS)
Changes in gut microbiome composition | Baseline & 4 days after
  To determine the changes of the composition and diversity of gut microbiome (genus & species) in faecal samples collected from participants via microbiome analysis after consumption of organic or non-organic plant-rich diet for 4 days

SECONDARY OUTCOMES:
Changes in flow-mediated-dilation (FMD) in the brachial artery | Baseline & 4 days after
  Determine changes in flow mediated dilation (FMD) of the brachial artery using a 12 MHz ultrasound transducer (Vivid I) coupled with a sphygmomanometer cuff after consumption of organic or non-organic plant-rich diet for 4 days
Changes in blood pressure | Baseline & 4 days after
  Determine changes in systolic and diastolic blood pressure after consumption of organic or non-organic plant-rich diet for 4 days
Changes in pulse wave velocity (PWV) | Baseline & 4 days after
  Determine changes in arterial stiffness via applanation tonometry after consumption of organic or non-organic plant-rich diet for 4 days. Carotid-femoral pulse wave velocity (cfPWV) will be measured using the SphygmoCor CvMS tonometer to produce PWV readings in m/s
Change in augmentation Index (AIx) | Baseline & 4 days after
  Determine the changes on augmentation Index (AIx) using a Sphygmocor device, after consumption of organic or non-organic plant-rich diet for 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rodriguez-Mateos, PhD, Principal Investigator — King's College London
Locations (1):
- Department of Nutritional Sciences, School of Life Course Sciences, Faculty of Life Sciences and Medicine, King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No